CLINICAL TRIAL: NCT06254391
Title: Very Low-dose Aspirin (30mg) vs. Standard Low-dose Aspirin (75mg) Among Patients Aged 65 Years or Above Undergoing PCI for Acute Coronary Syndrome: an Open-label Randomized Crossover Design Trial.
Brief Title: Aspirin Dose Comparison in Elderly PCI Patients: 30mg vs. 75mg in Acute Coronary Syndrome
Acronym: LowASA-PCI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Mariusz Tomaniak, Tomaniak Mariusz MD PhD Assoc. Prof., Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LowASA-PCI
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome
Keywords: Dual Antiplatelet Therapy; Myocardial Infarction; Acute Coronary Syndrome; Very-low dose aspirin; PCI
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: After collecting basic clinical information about the patients, patients undergoing percutaneous coronary intervention (PCI) due to acute coronary syndrome (within 24-48 hours after the procedure) will be randomized in a 1:1 scheme using the mobile application "Randomizer for Clinical Trial" (Medsharing, France) to one of the two arms of the study receiving ticagrelor at a maintenance dose of 90 mg twice daily, in which the following treatment sequence will be used (open-label crossover design):
  1. Aspirin (ASA) 30 mg once daily (morning) for 14 days followed by ASA 75 mg once daily (morning) for 14 days or
  2. ASA 75 mg once daily (morning) for 14 days, then ASA 30 mg once daily (morning) for 14 days.
  All patients will receive a loading dose of aspirin 300 mg before PCI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Very low-dose aspirin first (Other): Patients will receive ASA 30mg per day (in the morning) for 14 days, followed by ASA 75mg per day (in the morning) for the next 14 days.
  All the participants will receive standard maintenance dose of ticagrelor 90mg twice a day as part of the DAPT therapy. All the participants will receive the loading dose of ASA 300mg before the PCI procedure.
  Interventions: Drug: Low-dose aspirin
- Standard low-dose aspirin first (Other): Patients will receive ASA 75mg per day (in the morning) for 14 days, followed by ASA 30mg per day (in the morning) for the next 14 days.
  All the participants will receive standard maintenance dose of ticagrelor 90mg twice a day as part of the DAPT therapy. All the participants will receive the loading dose of ASA 300mg before the PCI procedure.
  Interventions: Drug: Low-dose aspirin

INTERVENTIONS:
Drug: Low-dose aspirin — Implementation of low-dose aspirin (30 mg)

SUMMARY:
Elderly patients undergoing percutaneous coronary intervention (PCI) face a high risk of both ischemic and hemorrhagic complications necessitating antiplatelet therapy. Previous data indicate that even at a dose of 20-30 mg/day, aspirin (ASA) allows almost complete inhibition of thromboxane (TX) A2 biosynthesis in healthy volunteers. However, ASA at a dose of 30 mg/day has not been evaluated in the acute phase of myocardial infarction or among elderly patients, where it may achieve an optimal balance between bleeding risk and ischemic complications.

This randomized study will include 40 patients over 65 years undergoing PCI for acute coronary syndrome (ACS). It compares a new dual antiplatelet therapy (DAPT) strategy consisting of a P2Y12 antagonist (ticagrelor) and ASA at a very low dose of 30 mg/day (n=20) against the current standard treatment (P2Y12 antagonist and ASA at a dose of 75 mg) (n=20) in the control group.

ELIGIBILITY:
Inclusion Criteria:

* age above 65 years
* acute coronary syndrome (ACS)
* positive results for myocardial necrosis markers (troponins)
* undergoing successful coronary angioplasty with stent implantation within the last 24-48 hours before enrollment in the study
* dual antiplatelet therapy (DAPT) containing ticagrelor

Exclusion Criteria:

* indications other than ACS and PCI for DAPT use
* history of stent thrombosis during the course of DAPT
* planned subsequent coronary artery revascularization
* planned surgery requiring suspension or interruption of DAPT
* planned discontinuation of ASA or P2Y12 antagonist during the study
* use of doses other than 75 mg ASA once daily or non-use of a P2Y12 inhibitor - intake of diuretic drugs (e.g., loop diuretics, thiazides, potassium-sparing drugs)
* intake or planned intake of oral anticoagulants, parenteral antithrombotic therapy (e.g., unfractionated heparin, low molecular weight heparin, bivalirudin), glycoprotein IIb/IIIa inhibitors (e.g., abciximab, tirofiban), fibrinolytic agents (e.g., tissue plasminogen activator), or nonsteroidal anti-inflammatory drugs
* history of acute or chronic liver disease; severe kidney disease requiring dialysis; pregnancy; comorbidities associated with a predicted life expectancy of less than 1 year
* any other condition deemed by the investigator to impact hemostasis, coagulation, bleeding risk, or the ability to adhere to the study protocol; receiving a strong inhibitor of cytochrome P450 3A, simvastatin or lovastatin at doses greater than 40 mg per day, a narrow therapeutic index cytochrome P450 3A substrate (e.g., cyclosporine or quinidine), or a strong inducer of cytochrome P450 3A (e.g., rifampin, rifabutin, phenytoin, carbamazepine, phenobarbital)
* hemodynamic instability; clinical condition preventing obtaining informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity (ASPI) | 14th day of treatment, 2h before ASA 30mg dose (through effect), and 2h after ASA 30mg dose (peak effect), in regards to group treated with DAPT with standard ASA 75mg dose after 14 days of therapy
  Comparison of platelet reactivity dependent on arachidonic acid (ASPI test) in low-dose ASA therapy, assessed in impedance aggregometry in regards to group treated with DAPT with standard ASA 75mg dose after 14 days of therapy.

SECONDARY OUTCOMES:
Platelet reactivity (ADP) | Days 7, 14, and 28 of treatment, 2 hours before the administration of the next ASA dose (pre-dose - representing the trough effect), and 2 hours after the ASA dose (post-dose - representing the peak effect)
  Comparison of platelet reactivity dependent on ADP (ADP test) in low-dose ASA therapy, assessed in impedance aggregometry in regards to the group treated with DAPT with standard ASA 75mg dose and level changes in individual patients.
Platelet reactivity (TRAP-6) | Days 7, 14, and 28 of treatment, 2 hours before the administration of the next ASA dose (pre-dose - representing the trough effect), and 2 hours after the ASA dose (post-dose - representing the peak effect)
  Comparison of platelet reactivity dependent on TRAP-6 protein activating the thrombin receptor (TRAP test) in low-dose ASA therapy, assessed in impedance aggregometry in regards to group treated with DAPT with standard ASA 75mg dose and level changes in individual patients.
Platelet reactivity (ASPI) | Days 7, and 28 of treatment, 2 hours before the administration of the next ASA dose (pre-dose - representing the trough effect), and 2 hours after the ASA dose (post-dose - representing the peak effect)
  Comparison of platelet reactivity dependent on arachidonic acid (ASPI test) in low-dose ASA therapy, assessed in impedance aggregometry in regards to group treated with DAPT with standard ASA 75mg dose and level changes in individual patients.
Bleeding time | Days 7, 14, and 28 of treatment 2 hours after the administration of the ASA dose
  Comparison of bleeding time (assessed with lancet method) between two groups (ASA 30mg and ASA 75mg) and among the individual patients.
PGI2 levels | Measured on days 7, 14, and 28 of treatment, 2 hours after the administration of the ASA dose
  Comparison of PGI2 concentration in urine between two groups (ASA 30mg and ASA 75mg) and among the individual patients.
TXB2 levels | Days 7, 14, and 28 of treatment, 2 hours before the administration of the next ASA dose, and 2 hours after the ASA dose
  Comparison of TXB2 concentration between two groups (ASA 30mg and ASA 75mg) and among the individual patients.

OTHER OUTCOMES:
Safety monitoring | 90th day
  Clinical endpoints (safety monitoring) will include an assessment of the composite endpoint comprising adverse cardiovascular events (MACE): death, myocardial infarction, stroke, and non-elective coronary artery revascularization within 3 months of PCI. The frequency of bleeding complications (BARC 1,2,3,4, or 5), and the frequency of confirmed and probable stent thrombosis defined by the Academic Research Consortium will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Mariusz Tomaniak, PhD, Principal Investigator — 1st Department and Clinic of Cardiology, Medical University of Warsaw
Locations (1):
- 1st Department and Clinic of Cardiology, Medical University of Warsaw, Warsaw, Mazowieckie Voivodenship, Poland

IPD SHARING:
Plan to Share IPD: No